CLINICAL TRIAL: NCT06102070
Title: Genetic Susceptibility to Severe Infections Including in Particular but Not Exhaustively All Types of Viral, Bacterialn and Fungal Infections.
Brief Title: Genetic Susceptibility to Severe Infections
Acronym: PREDISPOSITI
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C18-41
Record Dates: First submitted 2023-09-29; First posted 2023-10-26 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (10 ml) Skin biopsy (only for specific diseases as specified in the protocol) Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Predisposition: individuals suffering of having previously suffered of severe infectious diseases
  Interventions: Other: Blood samples drawing; Other: Skin biopsy

INTERVENTIONS:
Other: Blood samples drawing — 10 ml of periferal blood
Other: Skin biopsy — Skin biopsy only in some index cases depending of the pathology at the recruitment

SUMMARY:
Only a fraction of individuals infected with microbes develop clinical disease. This observation raises fundamental questions about the pathogenesis of infectious diseases. There is a complex interaction between environmental (microbial and non-microbial) and human (genetic and non-genetic) factors. This will determine the quality of the immune response against the infectious agent and the clinical manifestation. By definition, individuals who die from an infection have defective immunity to the pathogen in question (immune agent (immune deficiency).

The investigation of individual variability in the development of infectious diseases began in the early 20th. The first evidence to support the hypothesis that individual variability variability and immune deficiencies were hereditary came from observations of familial cases or genetic isolates genetic isolates (from a homogeneous population) of rare or common infectious diseases, which in some cases Mendelian heredity hat predisposition to infectious diseases runs in families even more so than diseases associated with less determined environmental factors, such as certain cancers. such as certain cancers. Finally, studies comparing the rate of concordance of infectious diseases between monozygotic and dizygotic twins also implicate genetic factors in disease susceptibility.

These observations were validated by the discovery of genetic defects associated with severe infectious diseases, leading to proof of concept. While a number of hereditary immune deficiencies associated with susceptibility to multiple pathogens or microorganisms, a growing number of new and rare new and rare immune deficiencies conferring restricted susceptibility to infections caused by a single caused by a single pathogen family, or even a single pathogen, in otherwise healthy children, have recently been identified (one gene, one pathogen). As a result, a dozen Mendelian clinical syndromes characterized by restricted susceptibility are now known. Over the last 20 years, it has been proven that these "idiopathic" infections were immune deficiencies.

The investigators now wish to study new severe infections, including but not limited to viral, fungal and bacterial infections. viral, fungal, bacterial and parasitic infections. This should lead to a better understanding of the pathophysiology of each disease, the development of new therapeutics and better patient care.

DETAILED DESCRIPTION:
Justification of the number of subjects:

The prevalence of the various severe infections we wish to explore ranges from one case in 50,000 to one case in 1,000,000 individuals; consequently, we plan to recruit only a small cohort of patients per pathology. Due to the exploratory nature of this research, no sample size calculation is possible.

ELIGIBILITY CRITERIA

Inclusion criteria :

1. Index cases (patients)

   * Informed consent signed by the patient. In the case of a minor patient, consent must be signed by the holders of parental authority. In the case of a protected adult patient, consent is signed by his or her signed by the patient's legal representative. In the case of an adult patient unable to consent at the time of consent is signed by a family member.
   * have a proven rare and severe infection defined by at least one of the following elements:

     * Acute, life-threatening infection requiring hospitalization, especially in an intensive particularly in intensive care.
     * Recurrent and/or chronic infections requiring frequent hospitalization or follow-up visits hospitalization or follow-up visits (dermatology, cardiology, neurology, infectious diseases, immunology, etc.), infectious diseases, immunology, etc.).
     * Acute and/or chronic infections leading to sequelae (motor or cognitive deficits, etc.).
     * Disseminated infection by an opportunistic microbe.
   * be hospitalized or followed in a specialized hospital ward, emergency room or intensive care unit
   * be affiliated to a Social Security scheme.
2. Related

   * have informed consent signed by the adult relative. In the case of a minor relative, the consent is consent is signed by the holders of parental authority. In the case of an adult relative the consent is signed by his or her legal representative
   * be related to the index case up to the 3rd degree: Parents, Children, Brother, Sister, Grandparents, Uncles, Aunts, Cousins, Nephews, Nieces
   * be affiliated to a Social Security system

Non-inclusion criteria :

1. Index case:4/4 C18-41 _Predisposition_Synopsis_V2.0_20220324

   * Acquired immunodeficiency (having received immunosuppressive treatment in the 3 months prior to the onset of the disease or HIV-positive)
   * Pregnant at the time of illness
   * Person under court protection
2. Related persons :

   * Pregnant or breast-feeding woman
   * Person under court protection

ELIGIBILITY:
Inclusion Criteria:

* to sign the informed consent signed by the patient. In the case of a minor patient, consent is signed by the holders of parental authority. In the case of a protected adult patient, the consent is signed by their legal representative. In the case of an adult patient unable to consent at the time of inclusion, consent is signed by a family member.
* to have a proven rare and severe infection
* to be hospitalized or followed in a specialized hospital department, in the emergency room or in intensive care
* to be affiliated to the French Social Security system
* for relatives, to be related to the index case up to the 3rd degree: Parents, Children, Brother, Sister, Grandparents, Uncles, Aunts, Cousins, Nephews, Nieces

Exclusion Criteria

* to have an acquired immunodeficiency (having received immunosuppressive treatment in the 3 months preceding the onset of the disease or being HIV positive)
* pregnant woman at the time of illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients (index cases) will be recruited on the basis of a proven diagnosis of severe infection, including in particular but not exhaustively severe viral, parasitic, fungal and/or bacterial infections, prospectively.
  2. Relatives of the applicant: Father, Mother, Brother, Sister, Grandparents, Uncles, Aunts, Cousins, Nephews, Nieces
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2037-02-17 (Estimated); Study Completion 2038-10-18 (Estimated)

PRIMARY OUTCOMES:
Identification of chromosomal regions associated with the disease through a "homozygosity mapping" study on multiplex and/or consanguineous families. | through study completion, an average of 10 years
  Whole genome genotyping using high density microarrays (Affymetrix 6.0 type or equivalent) on the gDNA of the index case and its relatives. Exome data will also be used for homozygosity calculation.
Identification of candidate genes for genetic susceptibility to infectious diseases | through study completion, an average of 10 years
  1. To sequence using the high-throughput sequencing technique (exome or genome).
  2. To check the genetic segregation of mutations identified in relatives in each family.
Validation of candidate genes as factor of susceptibility to infectious diseases | through study completion, an average of 10 years
  To validate the pathogenic effect of the mutation by functional and complementation tests on patient cells and control cells, and in an overexpression system

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Etudes des Déficits Immunitaires (CEDI), Hôpital Necker-Enfants, Paris, Île-de-France Region, France